CLINICAL TRIAL: NCT02750176
Title: Rehabilitation of Patients With Full-thickness Rotator Cuff Tears: Planning and Pilot Study for Feasibility and Efficacy
Brief Title: Rehabilitation: Closed-Chain Exercises for Rotator Cuff Tears
Acronym: CERCT
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Lori Michener, Professor, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-15-00771
Record Dates: First submitted 2016-04-18; First posted 2016-04-25 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Full Thickness Rotator Cuff Tear
Keywords: Rehabilitation; Closed chain exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CERCT (Experimental): Closed chain exercises
  Interventions: Other: Closed chain exercises

INTERVENTIONS:
Other: Closed chain exercises — Closed-chain strengthening will be performed with the shoulder moving over a fixed hand. Resistance will be provided by body weight against gravity. To off-load and progress the amount of body-weight resistance, elastic bands will be used to support body weight using a exercise frame. Patients will perform 6 exercises.

SUMMARY:
A single arm design will be used to assess the feasibility and preliminary efficacy of a closed-chain rehabilitation protocol for patients with full thickness rotator cuff tears of the shoulder. Full thickness rotator cuff tears will be documented using MRI or ultrasound images. 30 participants will be recruited for this study. The rehabilitation protocol will include two stages: stage 1, physical therapy, and stage 2, gym program. Stage I will include a total number of session between 12 and 24. The number of session included in stage 2, will depend on the total number of session completed during stage 1. The total duration of both stages will 5 months.

DETAILED DESCRIPTION:
Closed-chain exercises have been used extensively in rehabilitation approaches to treat a diverse range of musculoskeletal diagnoses. The closed-chain approach theoretically facilitates co-contraction to improve joint mobility, stability and motor control, as well as decreasing potential compression of the RC tendons in the subacromial space. The closed-chain exercises are performed with the hands in contact with the floor/table, while the shoulder joint moves and gravity provides resistance. This approach may prevent tear progression and improve joint mechanics, shoulder pain, and function.

STAGE 1 - Physical therapy

Participants will be provided closed-chain exercises in the physical therapy treatment by a licensed physical therapist. The length of each session will be 1 hour. Participants will attend 2 sessions per week, for a minimum of 12 sessions. The maximum number of sessions to complete Stage I of the protocol is 24. Each physical therapy session will consist of closed-chain strengthening, along with stretching and aerobic exercises.

During the closed-chain strengthening portion, participants will be asked to perform 6 exercises focusing on the shoulder girdle. Closed-chain strengthening will be performed with the shoulder moving over a fixed hand. Resistance will be provided by body weight against gravity. To off-load and progress the amount of body-weight resistance, elastic bands will be used to support body weight. The elastic bands will be attached to support frame used for the exercises. As the patient improves, less elastic band support will be provided to allow increased resistance via the patient's body weight. The criteria for determining if the resistance is too high or the exercise is too difficult will be based on 2 criteria: 1.) after the exercise is completed, the participant rates their shoulder pain > 2/10 increase as compared to baseline pain taken at the start of that day's treatment session, on the numeric pain rating scale, and 2.) BORG scale > 3 (moderate difficulty) and an inability of the participant to maintain proper exercise form and full range of motion. If these criteria are met then the physical therapist will modify the exercise so the subject can perform similar movement pattern without pain. The goal will be for the participant to perform 2 sets of 20 repetitions, of each exercise. When the participant is able to perform 24 repetitions with the given load, over 2 successive treatment sessions, then the resistance will be increased.

The investigators recognize that there is limited evidence regarding the effectiveness and safety of closed-chain exercises in patients with full-thickness rotator cuff tears. Therefore, the investigators are employing several steps to assure safety. At the beginning of each session, each patient will fill out a questionnaire to assess for adverse effects of exercises (such as severe joint pain). After each exercise, participants will rate their shoulder pain level and their perceived difficulty with the exercise. This information will be used to tailor the intervention according to the response to the intervention. Furthermore, it will allow for monitoring for adverse outcomes of the intervention.

Participants will perform aerobic exercises of a stationary bike, elliptical, and treadmill. Aerobic exercise will last about 10 to 15 minutes each session. Intensity of aerobic exercises will be adjusted throughout stage I. The target is to exercise at least at a 4 level (somewhat hard) on the BORG scale.

STAGE 2 - Gym program

Participants will be enrolled in a gym program following discharge from Stage 1. The Gym Program will be provided by a health care professionals trained in the delivery of exercise. Each session will be 1 hour. Participants will attend 2 sessions per week, for 8- 12 weeks depending on when they are discharged from Stage I. Each session will consist of closed-chain strengthening, stretching, and aerobic exercises.

During the closed-chain strengthening portion, participants will execute the same six-strengthening exercises as stage I. The next phase involves progressing to a moderate resistance load that will allow the participant to complete 2 sets of 8 to 12 repetitions of a given exercise. When the participant is able to perform more than 12 repetitions with a given load, over the course of 2 successive training sessions, then the resistance will be incrementally increased. The maximum resistance will be against body weight (no support from bands).

Participants will perform aerobic exercises alternating each session between a stationary bike, elliptical, and treadmill. Aerobic exercise will last about 15 to 20 minutes each session. Intensity of aerobic exercises will be adjusted throughout stage II. The target will be to exercise at least at a 4 level (somewhat hard) on the BORG scale.

ELIGIBILITY:
Inclusion Criteria:

* Full-thickness rotator cuff tears - confirmed by ultrasound (US) or magnetic resonance imagining (MRI)
* Symptomatic for > 3 months
* Reduction in shoulder function:

Patient satisfaction with use of their shoulder: ≤ 7/10 (10 = fully satisfied) OR Penn Function Subscale Score ≤ 40/60 (60 = full function)

Exclusion Criteria:

* Physical therapy for current shoulder symptoms within last 3 months
* Previous shoulder surgery on the involved shoulder
* Cervical radiculopathy
* Undergoing treatment for active cancer
* Cardiovascular, pulmonary, neurological disease with physician limitations on exercise
* Uncontrolled high blood pressure (> systolic above 90, diastolic above 140)
* Unstable shoulder - primary diagnosis
* Unable to complete up to 5 months of treatment at the clinic

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-04; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Feasibility - recruitment | End of the study (Stage 2): 5 months / approximately 24 weeks
  Recruit 65% of the patients with rotator cuff tears that come to the USC PT Associate clinic for physical therapy treatment or patients that are seen at the physician office and are referred for physical therapy treatment.
Patient Specific Functional Scale (PSFS) | End of the study (Stage 2): 5 months / approximately 24 weeks
Penn Shoulder Score (Penn) | End of the study (Stage 2): 5 months / approximately 24 weeks

SECONDARY OUTCOMES:
Feasibility - retention | End of the study (Stage 2): 5 months / approximately 24 weeks
  The goal is to retain at least 75% of the participants enrolled.
Quick Disabilities of the Arm Shoulder Hand (QDASH) scale | End of the study (Stage 2): 5 months / approximately 24 weeks
Global Rating of Change (GRoC) scale | End of the study (Stage 2): 5 months / approximately 24 weeks
Numeric Pain Rating Scale (NPRS) | End of the study (Stage 2): 5 months / approximately 24 weeks
American Shoulder and Elbow Surgeon Patient-report (ASES) scale | End of the study (Stage 2): 5 months / approximately 24 weeks
Shoulder pain-free active elevation range of motion | End of the study (Stage 2): 5 months / approximately 24 weeks
Shoulder elevation strength | End of the study (Stage 2): 5 months / approximately 24 weeks
Shoulder external rotation strength | End of the study (Stage 2): 5 months / approximately 24 weeks
Patient Acceptable Symptom State (PASS) score | End of the study (Stage 2): 5 months / approximately 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lori Michener, PT, ATC, PhD, Principal Investigator — University of Southern California
Locations (1):
- Clinical Biomechanics Orthopedic and Sports Outcomes Research Laboratory, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided